CLINICAL TRIAL: NCT04604236
Title: Increasing Family Engagement and Treatment Initiation Through Family Assessment, Motivation,and Linkage Intervention (FAMLI)
Brief Title: Family Assessment Motivation, and Linkage Intervention (FAMLI)
Acronym: FAMLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, DanicaKnight, Principal Investigator, Texas Christian University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA049079-01 (NIH)
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Mapping Enhanced Counseling (MEC); Active Linkage (AL)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mapping Enhanced Counseling (MEC) (Experimental): MEC will target attitudes and norms. Attitudes include motivation for change, such as problem recognition and a belief that treatment will help. Subjective norms include normative beliefs about SU in adolescence (e.g., belief that it is ok to allow SU with parental supervision; experimentation is normal) and expectations about treatment.
  Interventions: Behavioral: Mapping Enhanced Counseling
- Active Linkage (AL) (Experimental): AL will target perceived control. Perceived control includes perceived logistical barriers and the degree to which individuals feel they can overcome them.
  Interventions: Behavioral: Active Linkage

INTERVENTIONS:
Behavioral: Mapping Enhanced Counseling — Practitioner-led, collaborative discussion with the youth and their caregiver on co-creating guide maps for decision making around starting treatment and continuing substance use that can help users organize information and think through a series of steps, questions, and behavior choices. encountered when attempting to initiate substance use treatment services. MEC is a communication and decision-making approach that uses graphic visualization tools to train individuals to monitor and control their decision making, improve judgment and behavioral choices (self-regulation), and improve communication and mutual understanding.
  Arms: Mapping Enhanced Counseling (MEC)
Behavioral: Active Linkage — Practitioner-led, collaborative discussion with the youth and their caregiver on how to overcome barriers encountered when attempting to initiate substance use treatment services. Discussion focuses around the top barriers identified through assessment and identification of 1 or more treatment agency/options that fit the family's needs. Practitioner takes a more active role in addressing barriers to treatment by helping the family find ways to access resources for payment, childcare, or other needs, and actively linking them to the treatment provider (e.g., scheduling the initial appointment with family present).
  Arms: Active Linkage (AL)

SUMMARY:
The R34 study will integrate existing tools for use with JJ populations and examine the feasibility, acceptability, and preliminary efficacy of a caregiver-youth intervention aimed at increasing SU treatment initiation. The adaptive intervention incorporates three evidence-based components: 1) assessment of motivation and linkage-related barriers with personalized feedback, 2) Mapping-Enhanced Counseling (MEC) for improving readiness for change and interpersonal communication, and 3) Active Linkage (AL) for addressing logistical barriers to service initiation. Youth-caregiver dyads will be randomly assigned to receive an initial dose (2, 1-hr sessions) of either MEC or AL. After 30 days, participants will be classified as Responders (1 or more services initiated) or Non-responders (no service initiation). All participants will be randomized to one of two intervening interventions: an additional dose (2, 1-hr sessions) of the initial intervention (MEC or AL) or a different dose (2, 1-hr sessions of the other). The specific aims are to 1) integrate and adapt appropriate evidence-based intervention components as a dyadic intervention approach for JJ youth and caregivers; 2) test the feasibility, acceptability, and optimal configuration of the dyadic intervention components and the protocol used to evaluate effectiveness (including feasibility of recruitment, implementation, measurement); and 3) preliminarily explore a) whether an initial dose of MEC or AL is sufficient for promoting early initiation and engagement, b) whether an additional dose of MEC or AL or a change in dose is more effective, and c) which component sequence is most effective. Primary outcomes include youth (initiation of assessment or counseling; counseling attendance) and caregiver (attendance at assessment, first counseling, and/or family sessions) measures. Secondary outcomes include youth and caregiver attitudes (problem recognition, desire for help), normative beliefs (SU norms), perceived control (stressors and obstacles), and youth SU (self-report corroborated by UA results). The study addresses the sizeable gap in service receipt among JJ youth by addressing family engagement, and focuses on improving motivation to change, linkage to services, and treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* pre or post adjudicated or deferred prosecution
* have an identified SU need within the past 12 months (confirmed by the TCU Drug Screen-5 during initial assessment)
* speak English
* no indication of active suicide risk
* can identify one parent/guardian/responsible adult (caregiver) that is willing to participate who speaks Spanish or English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Youth Initiation | Week 4
  Youth attendance at 1 or more treatment appointment (assessment or counseling), obtained through self-report and corroborated using probation agency attendance records
Youth Initiation | Week 9
  Youth attendance at 1 or more treatment appointment (assessment or counseling), obtained through self-report and corroborated using probation agency attendance records
Youth Initiation | Week 17
  Youth attendance at 1 or more treatment appointment (assessment or counseling), obtained through self-report and corroborated using probation agency attendance records
Caregiver attendance with youth at 1 or more treatment appointment | Week 4
  Caregiver attendance with youth at 1 or more treatment appointment (assessment, counseling)
Caregiver attendance with youth at 1 or more treatment appointment | Week 9
  Caregiver attendance with youth at 1 or more treatment appointment (assessment, counseling)
Caregiver attendance with youth at 1 or more treatment appointment | Week 17
  Caregiver attendance with youth at 1 or more treatment appointment (assessment, counseling)

SECONDARY OUTCOMES:
Change in Youth Treatment Motivation as measured by the TCU MOT Form | Weeks 1, 9, and 17
  Change in motivation for treatment (problem recognition, desire for help, treatment readiness)
Change in Caregiver's Perception of Youth's Treatment Motivation as measured by the TCU MOT Form | Weeks 1, 9, and 17
  Change in motivation for treatment (recognition of youth's drug problem, desire for help, treatment readiness)
Change in Youth Normative Beliefs about Substance Use as measured by the TCU THK Form | Weeks 1, 9, and 17
  Change in beliefs about substance use (drug culture)
Change in Caregiver Normative Beliefs about Substance Use as measured by the TCU THK Form | Weeks 1, 9, and 17
  Change in beliefs about substance use (drug culture)
Change in Youth Perceived Control over Substance Use as measured by the TCU THK Form | Weeks 1, 9, and 17
  Change in perceived control over substance use
Change in Youth Perceived Control over Treatment Initiation as measured by the Barriers to Treatment Participation Scale (BTPS) | Weeks 1, 9, and 17
  Change in perceived control over treatment initiation (number of barriers to seeking and starting treatment)
Change in Caregiver Perceived Control over Youth's Substance Use as measured by the Caregiver Strain Questionnaire (CGSQ-SF7): | Weeks 1, 9, and 17
  Change in perceived control over youth's substance use (stressors and obstacles caused by youth's substance use)
Change in Caregiver Perceived Control over Youth's Treatment Initiation as measured by the Barriers to Treatment Participation Scale (BTPS) | Weeks 1, 9, and 17
  Change in perceived control over youth's treatment initiation (number of barriers to seeking and starting treatment)
Change in Youth Intentions to Use Substances as measured by the TCU THK Form | Weeks 1, 5, 9, and 17
  Change in intention to use substances (drug resistance efficacy) and to initiate treatment
Change in Youth Intentions to Initiate Treatment | Weeks 1, 5, 9, and 17
  Change in intention to initiate treatment
Change in Caregiver Intentions to schedule and attend youth's treatment sessions | Weeks 1, 5, 9, and 17
  Change in intention to initiate youth's substance use treatment (intention to contact agency, intention to accompany child)
Change in Youth Substance Use as measured by the TCUDS and Opioid Supplement Forms | Weeks 1, 5, 9, and 17
  Self-reported use of substances (e.g., alcohol, marijuana, opioids), corroborated by urinalysis
Change in Family relationships as measured by the TCU FFS Scale | Weeks 1, 9, and 17
  Change in quality of family relationships (warmth, control, conflict)
Change in Family responsiveness as measured by the Family Assessment Device (FAD) | Weeks 1, 9, and 17
  Change in quality of family affective responsiveness, affective involvement, behavior control)

CONTACTS AND LOCATIONS:
Overall Officials: Danica Knight, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No